CLINICAL TRIAL: NCT01120665
Title: Isolated and Associated Effects of Physical Exercise and Estrogen Therapy on Climactercs Women
Acronym: TRH01/989-7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Eduardo Moacyr Krieger, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TRH01/989-7
Record Dates: First submitted 2010-04-28; First posted 2010-05-11 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Women's Health
Keywords: women's health; hormone replacement therapy; exercise
MeSH Terms: conditions — Motor Activity | interventions — Estradiol; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PLACEBO-CONTROL (Experimental): PLACEBO + CONTROL TO EXERCISE
  Interventions: Drug: Placebo; Other: Control
- ESTROGEN THERAPY + CONTROL (Experimental): ESTROGEN THERAPY (estradiol valerate 1 mg/dia orally) + CONTROL TO EXERCISE
  Interventions: Drug: Estradiol valerate; Other: Control
- PLACEBO+AEROBIC TRAINING (Experimental): PLACEBO + AEROBIC TRAINING (cicle-ergometer, 50 minutes, 3x week)
  Interventions: Other: Aerobic training; Drug: Placebo
- ESTROGEN THERAPY + AEROBIC TRAINING (Experimental): ESTROGEN THERAPY (estradiol valerate 1 mg/dia orally) + AEROBIC TRAINING (cicle-ergometer, 50 minutes, 3x week)
  Interventions: Drug: Estradiol valerate; Other: Aerobic training

INTERVENTIONS:
Drug: Estradiol valerate — estradiol valerate, 1 mg/day, orally.
  Other Names: hormone therapy
  Arms: ESTROGEN THERAPY + AEROBIC TRAINING; ESTROGEN THERAPY + CONTROL
Other: Aerobic training — Aerobic trainin (cycleergometer, 3x/week, moderate intensity, 50 minutes)
  Other Names: physical training
  Arms: ESTROGEN THERAPY + AEROBIC TRAINING; PLACEBO+AEROBIC TRAINING
Drug: Placebo — lactose powder, corn starch, microcrystalline cellulose, and magnesium stearate
  Arms: PLACEBO+AEROBIC TRAINING; PLACEBO-CONTROL
Other: Control — The control group was advised to maintain their normal habits, and not to begin any physical exercise program during the study period
  Other Names: sedentary
  Arms: ESTROGEN THERAPY + CONTROL; PLACEBO-CONTROL

SUMMARY:
This study will investigate the isolated and the associated effect of estrogen therapy and physical exercise in the function, regulation and cardiovascular risk markers of 60 postmenopausal women, (45 - 60 years old). The volunteers will be randomaized into two groups: estrogen therapy (estradiol valerate 1 mg/day oraly) and placebo. The two groups will be randomaized into two subgroups: exercise group (aerobic trainning,cicle-ergometre, 50 minutes, 3 x week) and sedentary group. At 0, 6 and 12 months the volunteers will be submited to: clinical analise, cardiorespiratory analise (ergoepirometric test), quality of life questionare (Short Form-36 [SF-36]), ambulatory blood pressure monitoring during 24 hours and to 2 experimental sessions where the cardiovascular responses to insulin action (euglicemic/hiperinsulinemic clamp) and to physical and mental stress (microneurography) will be accessed. Besides these, the volunteers of the sedentary group will be submited to an extra session at 6 months of study evaluate the physiological answer to insulin infusion after an acute session of exercise.

DETAILED DESCRIPTION:
More than an isolated event, menopause is an universal process that produces many physiologic changes, affecting not only the reproductive tissues but other systems of women's body. Post-menopause period is usually accompanied by an increase in climacteric symptoms, which decrease healthy related quality of life. Moreover, many unhealthy changes occur at this period of women's life, increasing the risk for metabolic syndrome development, which might be due, at least in part, to an increase in insulin resistance and compensatory hyperinsulinemia.

Hormone therapy is indicated as the main treatment to reduce or relief the negative effects of menopause. Although many studies have confirmed the possible positive effects of this approach on postmenopausal symptoms, its effects on insulin resistance and other metabolic syndrome factors remain controversial.

On the other hand, it's well known that acute and chronic exercises can provide a wide range of benefits for postmenopausal women's health, including decrease of insulin resistance and symptoms relief.

In clinical practice, many postmenopausal women are using hormone therapy and are instructed to exercise. However, the effects of this association are poorly studied.

Thus, the main goal of this randomized placebo-controlled trial was to evaluate, in healthy, middle age, and hysterectomized postmenopausal women, the single and combined effects of physical exercise and oral estrogen use on blood pressure (BP), heart rate (HR), muscle blood flow, and autonomic function measured at baseline conditions and under hyperinsulinemia stimulus. Moreover, it also investigated the effects of these interventions on symptoms relief and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hysterectomy women, with or without ovaries, confirmed by transvaginal ultrasound.
* Climacteric women, postmenopausal for at least 1 year, with vasomotor symptoms (Kupperman, 1959) and/or laboratory diagnosis of menopause (high luteinizing hormone [LH] and follicle-stimulating hormone [FSH] and estradiol decreased).

Exclusion Criteria:

* Hypertension or other cardiovascular disease (thromboembolism, heart disease, myocardial infarction, stroke, vascular disorders, coronary insufficiency or venous)
* Osteoporosis.
* Diagnose or suspected breast cancer or ovaries.
* Current illness or a history of severe liver failure, jaundice or severe pruritus pregnancy and liver tumor.
* Endocrine and metabolic diseases as diabetes, thyroid disorders, obesity and dyslipidemia.
* Chronic diseases such as kidney diseases and collagen diseases.
* Women with cervical or vaginal malignancies.
* Hypersensitivity to estradiol valerate.
* Previous use of estrogen-containing implants in the last two years, use of hormone replacement therapy (HRT) orally or transdermally in the last three months or HRT use by injection in the last six months before the study start.
* Limited mobility or other physical problems that contraindicate the physical exercises.
* Women who are engaged in regular physical activity.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2002-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure | six months
  Blood pressure will be measured as often as needed, respecting the interval 1-2 minutes among measurements, until you obtain three consecutive measurements with a difference of less than 5 mmHg by auscultation and oscilometric methods. The verification of calibration of the monitor is often assessed by comparison with the mercury.

SECONDARY OUTCOMES:
hemodynamics mechanisms | six months
  Hemodynamics mechanisms will be evaluate by air-occlusion pletismography
autonomics mechanisms | six months
  autonomics mechanisms will be evaluated by microneurography methods and heart rate and blood pressure variability

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Fonseca, PhD, Principal Investigator — University of Sao Paulo; Decio Mion Jr, PhD, Principal Investigator — University of Sao Paulo; Claudia LM Forjaz, PhD, Principal Investigator — University of Sao Paulo; Sandra B Abrahão, PhD, Principal Investigator — University of Sao Paulo; Taís Tinucci, PhD, Principal Investigator — University of Sao Paulo